CLINICAL TRIAL: NCT02231866
Title: VRC 207: A Phase I/1b, Open-Label, Dose-Escalation Clinical Trial to Evaluate the Safety, Tolerability and Immunogenicity of the Ebola Chimpanzee Adenovirus Vector Vaccines, VRC-EBOADC069-00-VP (cAd3-EBO) and VRC-EBOADC076-00-VP (cAd3-EBOZ), in Healthy Adults
Brief Title: Safety, Tolerability, and Immunogenicity of the Ebola Chimpanzee Adenovirus Vector Vaccine (cAd3-EBO), VRC-EBOADC069-00-VP, in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 140183; 14-I-0183
Record Dates: First submitted 2014-09-03; First posted 2014-09-04 (Estimated); Last update posted 2018-07-05 (Actual); Status verified 2017-04-05

CONDITIONS: Healthy Adult Immune Responses to Vaccine
Keywords: Filovirus; Healthy; Ebola Hemorrhagic Fever; Immunity; Ebola Virus
MeSH Terms: conditions — Hemorrhagic Fever, Ebola

ARMS (6):
- Group 1 (Experimental): cAd3-EBO at 2x10(10)PU IM
  Interventions: Biological: VRC-EBOADC069-00-VP
- Group 2 (Experimental): cAd3-EBO at 2x10(11)PU IM
  Interventions: Biological: VRC-EBOADC069-00-VP
- Group 3 (Experimental): cAd3-EBO at 2x10(11)PU IM boost of Ebola DNA WT vaccine (VRC 206 participants)
  Interventions: Biological: VRC-EBOADC069-00-VP
- Group 4A (Experimental): cAd3-EBOZ at 1x10(10)PU IM
  Interventions: Biological: VRC-EBOADC076-00-VP
- Group 4B (Experimental): cAd3-EBOZ at 1x10(11)PU IM
  Interventions: Biological: VRC-EBOADC076-00-VP
- Group 5 (Experimental): cAd3-EBO at 2x10(11)PU IM
  Interventions: Biological: VRC-EBOADC069-00-VP

INTERVENTIONS:
Biological: VRC-EBOADC069-00-VP — cAd3-EBO Ebola Chimpanzee Adenovirus Vector Vaccine GP Zaire + GP Sudan
  Arms: Group 1; Group 2; Group 3; Group 5
Biological: VRC-EBOADC076-00-VP — cAd3-EBO Ebola Chimpanzee Adenovirus Vector Vaccine GP Zaire
  Arms: Group 4A; Group 4B

SUMMARY:
Background:

- Ebola virus causes an infection known as Ebola virus disease (EVD). This it is generally a severe disease which can also lead to death. The 2014 outbreak of EVD in West Africa is the largest ever. Researchers want to develop a vaccine to prevent Ebola infection. It is impossible for someone to get an Ebola infection from this vaccine.

Objectives:

- To see if an Ebola vaccine is safe and to study immune responses to it.

Eligibility:

- Healthy adults ages 18-65.

Design:

* Participants will be screened through a separate protocol.
* Participants will receive the vaccine injection by needle and syringe into an upper arm muscle. - Participants will stay at the clinic for 3 hours after the injection.
* About 2 days later, participants must speak with clinic staff about how they are doing.
* Every day for 7 days after the injection, participants will record their temperature and symptoms and look at the injection site. They will get a thermometer and a ruler to measure any redness or swelling. They will report any side effects.
* In the first 2 months in the study, participants will have at least 6 clinic visits and 1 phone call. They will have at least 3 other visits over the next 9 months.
* At each visit, participants will be checked for health changes or problems since their last visit. They will be asked how they feel and if they have taken any medicine. Blood will be drawn at most visits. Urine samples may be collected.

DETAILED DESCRIPTION:
Study Design: This is a Phase 1/1b, open-label study to examine safety, tolerability and immunogenicity of investigational Ebola vaccines in healthy adults. Part 1 is a Phase 1 dose escalation of the cAd3-EBO vaccine that encodes wild type (WT) glycoproteins (GP) from Zaire and Sudan strains of Ebolavirus. Part 2 is a Phase 1b further evaluation of the cAd3-EBO vaccine at the highest dose and evaluation of the Zaire component, which will be provided as a vaccine designated cAd3-EBOZ. The hypotheses are that the study vaccines, cAd3-EBO and cAd3-EBOZ, will be safe and will elicit immune responses to Ebola GP. The primary objectives are to evaluate the safety and tolerability of the study vaccines administered as single intramuscular (IM) injections at two dose levels. The secondary objectives are related to evaluation of the immunogenicity.

Product Description: VRC-EBOADC069-00-VP (cAd3-EBO) is composed of two recombinant cAd3 vectors in a 1:1 ratio that express Ebola WT GPs from Zaire and Sudan strains. It is formulated at 2 times 10(11) PU/mL.

VRC-EBOADC076-00-VP (cAd3-EBOZ) is composed of a cAd3 vector that expresses Ebola WT GP from the Zaire strain. It is formulated at 1 times 10(11) PU/mL.

VRC-DILADC065-00-VP (diluent) is the formulation buffer used for vaccine production and will be used when needed to prepare the correct dosage of cAd3-EBO and cAd3-EBOZ.

Subjects: Part 1: Healthy adult volunteers, 18 to 50 years old;

Part 2: Healthy adult volunteers, 18 to 65 years old.

Study Plan: Part 1: 20 subjects will be enrolled, with 10 in each of the two dosage groups for cAd3-EBO. The dose escalation plan includes daily review of any new safety data by a study clinician, weekly review of safety data by the protocol team and a staged enrollment plan with required interim safety reviews before proceeding to the next step. The study plan includes no more than one enrollment per day for the first 3 vaccinated subjects in each group. After at least 3 days of follow-up, an interim safety review will occur before enrollment of additional subjects into the group. When there are at least 2 weeks of follow-up safety data for the first 3 vaccinated subjects in Group 1, an interim safety review will occur before proceeding to the next dose level.

Part 2: About 130 subjects will be enrolled as shown in the Schema table.

Group 3 is open only to subjects who received Ebola DNA WT vaccine in protocol VRC 206 to receive cAd3-EBO as a booster vaccine at the 2 times 10(11) PU dose.

Group 4 is for randomization of subjects to two dosage groups of cAd3-EBOZ.

Group 5 is for further evaluation of the cAd3-EBO vaccine at the 2 times 10(11) PU dose.

Study Duration: Subjects will be evaluated by 9 clinic visits over 48 weeks.

ELIGIBILITY:
* INCLUSION CRITERIA:

A volunteer must meet all of the following criteria:

1. 18 to 50 years old for Groups 1 and 2; 18 to 65 years old for Groups 3, 4, and 5.
2. Available for clinical follow-up through Week 48 after enrollment for groups 1-4 and through at least Week 4 after enrollment for group 5, with no planned travel that would preclude completion of the Study Week 4 visit.
3. Able to provide proof of identity to the satisfaction of the study clinician completing the enrollment process.
4. Able and willing to complete the informed consent process.
5. Willing to donate blood for sample storage to be used for future research.
6. In good general health without clinically significant medical history.
7. Physical examination and laboratory results without clinically significant findings and a body mass index (BMI) less than or equal to 40 within the 56 days prior to enrollment.
8. For Group 3 volunteers only, must have received the VRC-EBODNA023-00-VP (Ebola DNA WT) vaccine in the VRC 206 study.

   Laboratory Criteria within 56 days prior to enrollment:
9. Hemoglobin greater than or equal to 11.5 g/dL for women; greater than or equal to 13.0 g/dL for men.
10. White blood cells (WBC) = 3,300-12,000 cells/mm(3).
11. WBC differential either within institutional normal range or accompanied by the Principal Investigator (PI) or designee approval.
12. Total lymphocyte count greater than or equal to 800 cells/mm(3).
13. Platelets = 125,000 400,000/mm(3).
14. Alanine aminotransferase (ALT) less than or equal to 1.25 times upper limit of normal.
15. Serum creatinine less than or equal to 1 times upper limit of normal.
16. Partial thromboplastin time (PTT) within institutional normal range.
17. Prothrombin time (PT) within institutional normal range or accompanied by the Principal Investigator (PI) or designee approval.
18. HIV-uninfected as evidenced by a negative FDA-approved HIV diagnostic blood test.

    Female-Specific Criteria:
19. Negative Beta-HCG (human chorionic gonadotropin) pregnancy test (urine or serum) on day of enrollment if woman is presumed to be of reproductive potential.
20. Agrees to use an effective means of birth control from at least 21 days prior to enrollment through 24 weeks after study vaccination if presumed to be of reproductive potential.

EXCLUSION CRITERIA:

A volunteer will be excluded if one or more of the following conditions apply:

Volunteer has received any of the following substances:

1. Investigational Ebola or Marburg vaccine in a prior clinical trial (except for Group 3 volunteers) or prior receipt of a cAd3 adenoviral vectored investigational vaccine.
2. Immunosuppressive medications within 2 weeks prior to enrollment.
3. Blood products within 112 days (16 weeks) prior to enrollment.
4. Investigational research agents within 28 days (4 weeks) prior to enrollment.
5. Live attenuated vaccines within 28 days (4 weeks) prior to enrollment.
6. Subunit or killed vaccines within 14 days (2 weeks) prior to enrollment.
7. Current anti-tuberculosis prophylaxis or therapy.

   Female-specific criteria:
8. Woman who is breast-feeding or planning to become pregnant during the first 24 weeks after study vaccine administration.

   Volunteer has a history of any of the following clinically significant conditions:
9. Serious adverse reactions to vaccines such as anaphylaxis, urticaria (hives), respiratory difficulty, angioedema, or abdominal pain.
10. Clinically significant autoimmune disease or immunodeficiency.
11. Asthma that is not well controlled.
12. Diabetes mellitus (type I or II), with the exception of gestational diabetes.
13. Thyroid disease that is not well controlled.
14. A history of hereditary angioedema (HAE), acquired angioedema (AAE), or idiopathic forms of angioedema.
15. Idiopathic urticaria within the last 1 year.
16. Hypertension that is not well controlled.
17. Bleeding disorder diagnosed by a doctor (e.g. factor deficiency, coagulopathy, or platelet disorder requiring special precautions) or significant bruising or bleeding difficulties with IM injections or blood draws.
18. Malignancy that is active or history of a malignancy that is likely to recur during the period of the study.
19. Seizure in the past 3 years or treatment for seizure disorder in the past 3 years.
20. Asplenia or functional asplenia.
21. Psychiatric condition that precludes compliance with the protocol; past or present psychoses; or within five years prior to enrollment, history of a suicide plan or attempt.
22. Any medical, psychiatric, social condition, occupational reason or other responsibility that, in the judgment of the investigator, is a contraindication to protocol participation or impairs a volunteer s ability to give informed consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2014-08-27; Primary Completion 2017-04-05 (Actual); Study Completion 2017-04-05 (Actual)

PRIMARY OUTCOMES:
Solicited systemic and local reactogenicity signs and symptoms. | Daily for 7 days following each vaccination.
Occurrence of adverse events of all severities. | Through 4 weeks after the vaccination.
Occurrence of serious adverse events and new chronic medical conditions. | Through 48 weeks after the vaccination.

SECONDARY OUTCOMES:
Antibody responses as measured by ELISA and neutralization assays | 4 weeks after vaccination
T cell immune responses as measure by intracellular cytokine staining (ICS) | 4 weeks after vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Julie E Ledgerwood, D.O., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (3):
- United States (3):
  - Hope Clinic - Emory Vaccine Ctr, Decatur, Georgia
  - University of Maryland Center for Vaccine Development, Baltimore, Maryland
  - National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland

REFERENCES:
- [Background] Ledgerwood JE, Costner P, Desai N, Holman L, Enama ME, Yamshchikov G, Mulangu S, Hu Z, Andrews CA, Sheets RA, Koup RA, Roederer M, Bailer R, Mascola JR, Pau MG, Sullivan NJ, Goudsmit J, Nabel GJ, Graham BS; VRC 205 Study Team. A replication defective recombinant Ad5 vaccine expressing Ebola virus GP is safe and immunogenic in healthy adults. Vaccine. 2010 Dec 16;29(2):304-13. doi: 10.1016/j.vaccine.2010.10.037. Epub 2010 Oct 27. PMID 21034824
- [Background] Martin JE, Sullivan NJ, Enama ME, Gordon IJ, Roederer M, Koup RA, Bailer RT, Chakrabarti BK, Bailey MA, Gomez PL, Andrews CA, Moodie Z, Gu L, Stein JA, Nabel GJ, Graham BS. A DNA vaccine for Ebola virus is safe and immunogenic in a phase I clinical trial. Clin Vaccine Immunol. 2006 Nov;13(11):1267-77. doi: 10.1128/CVI.00162-06. Epub 2006 Sep 20. PMID 16988008
- [Background] Kuhn JH, Bao Y, Bavari S, Becker S, Bradfute S, Brister JR, Bukreyev AA, Chandran K, Davey RA, Dolnik O, Dye JM, Enterlein S, Hensley LE, Honko AN, Jahrling PB, Johnson KM, Kobinger G, Leroy EM, Lever MS, Muhlberger E, Netesov SV, Olinger GG, Palacios G, Patterson JL, Paweska JT, Pitt L, Radoshitzky SR, Saphire EO, Smither SJ, Swanepoel R, Towner JS, van der Groen G, Volchkov VE, Wahl-Jensen V, Warren TK, Weidmann M, Nichol ST. Virus nomenclature below the species level: a standardized nomenclature for natural variants of viruses assigned to the family Filoviridae. Arch Virol. 2013 Jan;158(1):301-11. doi: 10.1007/s00705-012-1454-0. Epub 2012 Sep 23. PMID 23001720
- [Derived] Tapia MD, Sow SO, Lyke KE, Haidara FC, Diallo F, Doumbia M, Traore A, Coulibaly F, Kodio M, Onwuchekwa U, Sztein MB, Wahid R, Campbell JD, Kieny MP, Moorthy V, Imoukhuede EB, Rampling T, Roman F, De Ryck I, Bellamy AR, Dally L, Mbaya OT, Ploquin A, Zhou Y, Stanley DA, Bailer R, Koup RA, Roederer M, Ledgerwood J, Hill AVS, Ballou WR, Sullivan N, Graham B, Levine MM. Use of ChAd3-EBO-Z Ebola virus vaccine in Malian and US adults, and boosting of Malian adults with MVA-BN-Filo: a phase 1, single-blind, randomised trial, a phase 1b, open-label and double-blind, dose-escalation trial, and a nested, randomised, double-blind, placebo-controlled trial. Lancet Infect Dis. 2016 Jan;16(1):31-42. doi: 10.1016/S1473-3099(15)00362-X. Epub 2015 Nov 4. PMID 26546548
- [Derived] Ledgerwood JE, DeZure AD, Stanley DA, Coates EE, Novik L, Enama ME, Berkowitz NM, Hu Z, Joshi G, Ploquin A, Sitar S, Gordon IJ, Plummer SA, Holman LA, Hendel CS, Yamshchikov G, Roman F, Nicosia A, Colloca S, Cortese R, Bailer RT, Schwartz RM, Roederer M, Mascola JR, Koup RA, Sullivan NJ, Graham BS; VRC 207 Study Team. Chimpanzee Adenovirus Vector Ebola Vaccine. N Engl J Med. 2017 Mar 9;376(10):928-938. doi: 10.1056/NEJMoa1410863. Epub 2014 Nov 26. PMID 25426834